CLINICAL TRIAL: NCT02727543
Title: Medication Adherence Improvement Support App For Engagement - Blood Pressure
Acronym: MedISAFE-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Medisafe, Inc. (Industry); Evidation Health (Industry)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School and Executive Director, Center for Healthcare Delivery Sciences, Department of Medicine, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00015278
Record Dates: First submitted 2016-03-31; First posted 2016-04-04 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Hypertension; mHealth; Medication Non-adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants randomized to this arm will not receive the intervention.
- Intervention (Experimental): Participants randomized to this arm will receive the intervention, Medisafe, a smartphone application.
  Interventions: Other: Medisafe

INTERVENTIONS:
Other: Medisafe — Medisafe is a smartphone application available to download for free on any iOS or Android device. Medisafe addresses non-adherence by providing alerts to patients when it is time to take their medications. Other features include the ability to allow a "Medfriend" to check in if a medication is not taken, weekly reports of medication adherence, and monitoring of biometric measurements
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the impact of the Medisafe smartphone application on blood pressure control and self-reported medication adherence for patients with uncontrolled blood pressure.

DETAILED DESCRIPTION:
The Medication adherence Improvement Support App For Engagement - Blood Pressure (MEDISAFE-BP) trial is a prospective, intent-to-treat randomized control trial that will evaluate the impact of the Medisafe smartphone application on blood pressure control and self-reported medication adherence for patients with uncontrolled blood pressure.

Recruitment will be conducted by Evidation Health, which uses an online strategy to virtually announce, recruit, verify eligibility and enroll participants in clinical studies. Potential study subjects will be evaluated for inclusion and exclusion criteria, will give informed consent, complete the baseline assessment, and then be sent a Bluetooth-enabled home blood pressure cuff to verify that they have uncontrolled blood pressure (systolic blood pressure ≥ 140 mmHg but overall blood pressure ≤ 180/120 mmHg). Patients will be provided with a study overview and blood pressure measurement guide that will outline how to set up the monitor and take an accurate measurement, as well as the standard insert for how to use the home monitor and its associated smartphone application. Blood pressure readings will be electronically transmitted to Evidation Health via an Application Program Interface (API) with the blood pressure monitor manufacturer. Blood pressure will be calculated as the average of two measurements that are taken five minutes apart. Once their blood pressure readings have been confirmed as being elevated, patients will undergo randomization in a 1:1 ratio to intervention or control using simple randomization through a random number generated at the time of study enrollment.

Analyses will be performed by an intent-to-treat basis, where subjects will be analyzed in the groups they are assigned to during randomization. We will use linear regression to assess the impact of Medisafe on the study's two primary outcomes (change in systolic blood pressure and self-reported adherence) between the two study groups, three months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 75 years of age
* Self-reported systolic blood pressure greater than or equal to 140 mmHg
* Self-reported use of 1-3 of the following anti-hypertensive medications (thiazide, CCB, beta-blocker, ACE-I, ARB)
* Systolic blood pressure greater than or equal to140 mmHg (+/- diastolic blood pressure greater than or equal to 90 mmHg), but blood pressure less than or equal to 180/120 mmHg confirmed by home BP-cuff

Exclusion Criteria:

* Current use of a smartphone medication adherence application
* No ownership of a smartphone with iOS or Android operating system
* Currently taking more than 3 anti-hypertensive medications (thiazide, CCB, beta-blocker, ACE-I, ARB) by self report
* Currently undergoing dialysis
* Currently receiving chemotherapy or radiation
* Does not understand English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Three months after randomization
Self-reported medication adherence | Three months after randomization

SECONDARY OUTCOMES:
Change in number of subjects who have well controlled blood pressure | Three months after randomization
  Well controlled blood pressure <140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Center for Healthcare Delivery Sciences, Brigham and Women's Hospital
Locations (1):
- Evidation Health, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morawski K, Ghazinouri R, Krumme A, Lauffenburger JC, Lu Z, Durfee E, Oley L, Lee J, Mohta N, Haff N, Juusola JL, Choudhry NK. Association of a Smartphone Application With Medication Adherence and Blood Pressure Control: The MedISAFE-BP Randomized Clinical Trial. JAMA Intern Med. 2018 Jun 1;178(6):802-809. doi: 10.1001/jamainternmed.2018.0447. PMID 29710289